CLINICAL TRIAL: NCT01275599
Title: A Phase 1, Open-Label, Single-Sequence Study to Examine the Effect of Telaprevir on the Pharmacokinetics of Buprenorphine in Subjects on Stable Buprenorphine/Naloxone Maintenance Therapy
Brief Title: Drug-Drug Interaction Study Between Telaprevir and Buprenorphine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Tibotec BVBA (Industry)
Responsible Party: Scott McCallister, M.D., Vertex Pharmaceuticals Incorporated
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX10-950-024
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Hepatitis C; Opioid-Related Disorders
MeSH Terms: conditions — Hepatitis C; Opioid-Related Disorders | interventions — telaprevir; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label Arm (Experimental): The treatment period will include 3 phases:
  * 14 day run-in period
  * 7 day co-administration period
  * 31 day follow-up period
  Interventions: Drug: telaprevir; Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: telaprevir — Two 375 mg tablets administered every 8 hours on Day 1 through Day 7, inclusive.
Drug: buprenorphine/naloxone — Buprenorphine/naloxone sublingual tablets or films contain buprenorphine HCl and naloxone HCl dihydrate at a ratio of 4:1 buprenorphine:naloxone (ratio of free bases). In this study buprenorphine/naloxone will be dosed from Day -14 through Day 38, inclusive. From Day -14 through Day -1 all subjects will receive a maximum of 24 mg/6 mg of buprenorphine/naloxone. Subjects will not be permitted to change their dose during the telaprevir co-administration period (Day 1 through Day 7) unless warranted by the investigator's clinical judgment of subject safety. After Day 8, the dose of buprenorphine/naloxone may be adjusted if deemed necessary by the investigator.
  Other Names: Suboxone

SUMMARY:
The purpose of this study is to investigate the drug-drug interaction potential between telaprevir and buprenorphine/naloxone. An understanding of the interaction potential will help to determine whether buprenorphine dose adjustments are necessary for patients who are concomitantly treated with telaprevir.

Telaprevir, in combination with other antiviral agents, is being investigated for the treatment of chronic hepatitis C virus infection. Buprenorphine/naloxone is used for maintainance therapy in patients with opioid dependence.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 64 years, inclusive. Females must be of non-childbearing potential.
* Receiving once daily buprenorphine/naloxone maintenance therapy at a stable dose not exceeding 24 mg/6 mg, respectively, for at least 2 weeks prior to screening.

Exclusion Criteria:

* Illicit use of drugs such as cocaine, amphetamines and methylenedioxymethamphetamine (MDMA), barbiturates, benzodiazepines, tricyclic antidepressants, methadone or opiates/opioids (apart from buprenorphine).
* Treatment with any investigational drug within the last 30 days, or 5 half-lives, whichever is longer.
* Blood donation of 500 mL or more within the last 56 days.
* Infected with hepatitis B virus, hepatitis C virus, or human immunodeficiency virus (HIV).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Blood levels of buprenorphine | Day -4 through Day 38
  Measured by maximum observed concentration (Cmax), minimum observed concentration (Cmin), time of the maximum concentration (tmax), area under the time curve (AUC) from the time of study drug administration, zero to tau, where tau is the dosing interval.
Blood levels of norbuprenorphine | Day -4 through Day 38
  Measured by maximum observed concentration (Cmax), minimum observed concentration (Cmin), time of the maximum concentration (tmax), area under the time curve (AUC) from the time of study drug administration, zero to tau, where tau is the dosing interval.
Blood levels of naloxone | Day -1 and Day 7
  Measured by maximum observed concentration (Cmax)
Blood levels of telaprevir | Day 1 through Day 7
  Measured by maximum observed concentration (Cmax), minimum observed concentration (Cmin), time of the maximum concentration (tmax), area under the time curve (AUC) from the time of study drug administration, zero to tau, where tau is the dosing interval.

SECONDARY OUTCOMES:
Safety and tolerability | Day -14 through Day 38
  Measured by incidence of treatment-emergent adverse events, clinical laboratory assessments, electrocardiogram outcomes, and vital signs.
Buprenorphine withdrawal symtoms | Day -2 through Day 38
  Measured by Clinical Opiate Withdrawal Scale (COWS), Desires for Drug Questionnaire (DDQ), and pupillometry.

CONTACTS AND LOCATIONS:
Overall Officials: Scott McCallister, M.D., Study Director — Vertex Pharmaceuticals Incorporated
Locations (2):
- United States (2):
  - Overland Park, Kansas
  - Salt Lake City, Utah